CLINICAL TRIAL: NCT04633434
Title: Utilizing Smart Speaker Technology to Deliver Parenting Education Support to Parents of Young Children
Brief Title: Evaluation Study of Talk Parenting Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HD101190; R43HD101190-01A1 (NIH)
Record Dates: First submitted 2020-10-28; First posted 2020-11-18 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Parenting Practices; Self Efficacy; Stress; Child Behavior; Emotional Adjustment; Sleep Problems; Parent-Child Relations
Keywords: Feasibility; Satisfaction; Usability
MeSH Terms: conditions — Child Behavior; Parasomnias; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Behavioral (e.g., Psychotherapy, Lifestyle Counseling) In a 4-week period, families use at home a prototype Bedtime Routine module of the Talk Parenting program, a smart speaker app designed to provide parents with in-situ experiential support for building positive family routines. The prototype Bedtime Routine module of Talk Parenting guides families in creating a healthy bedtime routine to foster healthy sleep habits, provide experiential practice in self-regulation skills, and promote a positive parent-child relationship.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Talk Parenting Skill for Alexa - Parent (Experimental): 49 parents will be assessed at enrollment, then provided an Amazon Echo Dot and exposed to the prototype Bedtime Routine module of the Talk Parenting program for 4 weeks, and then re-assessed at 4 weeks (at treatment completion)
  Interventions: Behavioral: The Talk Parenting Skill for Alexa
- The Talk Parenting Skill for Alexa - Child (Experimental): Although 49 children were considered enrolled participants that actively participate in the intervention, we obtained no assessment data from the children themselves.
  Interventions: Behavioral: The Talk Parenting Skill for Alexa

INTERVENTIONS:
Behavioral: The Talk Parenting Skill for Alexa — In a 4-week period, families use at home a prototype Bedtime Routine module of the Talk Parenting program, a smart speaker app designed to provide parents with in-situ experiential support for building positive family routines. The prototype Bedtime Routine module of Talk Parenting guides families in creating a healthy bedtime routine to foster healthy sleep habits, provide experiential practice in self-regulation skills, and promote a positive parent-child relationship.

SUMMARY:
After development of the prototype Bedtime Routine module of the Talk Parenting program, the investigators will evaluate its feasibility and initial efficacy in a within-subjects pre-post design study. Through recruitment partner agencies, the investigators will recruit a sample of 49 at-risk families (49 primary parents, 49 target children). Primary parents will be assessed at enrollment via online an questionnaire, then provided an Amazon Echo Dot and asked to use the Bedtime Routine module for 4 weeks. They will then be re-assessed with the online questionnaire at 4 weeks (at treatment completion). Although children were considered enrolled participants that actively participate in the intervention, we obtained no assessment data from the children themselves.

DETAILED DESCRIPTION:
Parents provide consent for their own participation, as well as the participation of their target child (their child aged 3-5 years who presents the most behavioral challenges). After consent, primary parents complete the baseline (T1) questionnaire via the Qualtrics online assessment platform and then are provided an Echo Dot with the Bedtime Routine module enabled. After 4 weeks post-baseline, they are administered the T2 questionnaire. This design allows evaluation of T1-T2 change and satisfaction/usability of the Bedtime Routine prototype module. Although children were considered enrolled participants that actively participate in the intervention, we obtained no assessment data from the children themselves.

T1 and T2 questionnaires measure primary parents' parenting practices, self-efficacy, and stress; children's behavior, emotional adjustment, and sleep problems; and the parent-child relationship. The T2 questionnaire also contains measures of parent satisfaction, acceptability, and usability of the Talk Parenting skill, as well as any difficulties experienced, or problems made worse. Demographics are collected at T1. T1 and T2 questionnaires are administered via Qualtrics, an online assessment tool. Project staff follow-up with parents as needed to encourage questionnaire completion in a timely manner. Parents are paid $20 per assessment.

Families are provided an Echo Dot device with the Talk Parenting skill already enabled using a research Amazon account created for each family. The Echo Dot devices are paired with portable auxiliary battery packs to enable mobile use within the home, so that the device can be carried from room to room during execution of the bedtime routine. The devices are preconfigured by project staff onto research Amazon accounts. All families are provided a pre-configured wifi adaptor that creates a wifi network specific for the Echo Dot device to connect to. After the baseline assessment (T1), primary parents are mailed their Echo Dot device, portable auxiliary battery pack, wifi adaptor, and set-up instructions; staff provide follow-up phone support as needed. Usage data show whether families have used the device; project staff contact the parents to assist set up if parents have not enabled/used the device within 2 weeks. To ensure exposure to Talk Parenting, parents are asked to engage with the skill at least twice per week (or at least eight times); project staff prompt parents two to three times (via text, email, or phone, depending on parents' preference) during the 4-week period to encourage usage and provide technical support as needed.

At the end of the study, families are asked to return the wifi adaptor to the project offices; families are free to keep the Echo Dot device and auxiliary battery pack.

ELIGIBILITY:
Inclusion:

1. Parent learned about the study through a participating agency
2. Child 3-5 years old who lives with the parent at least half time
3. Parent puts the child to bed at least 2 nights per week
4. Able to read and understand English
5. Has access to the internet at home.

Exclusion:

1. Families of target-age children with a developmental disability severe enough that the child cannot speak or follow simple directions will be excluded; their needs are beyond the scope of Talk Parenting.

Ages: 3 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Smith, Ph.D., Principal Investigator — Oregon Research Behavioral Interventions Strategies, Inc.
Locations (1):
- David R Smith, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berry JO, Jones WH. The Parental Stress Scale: Initial Psychometric Evidence. Journal of Social and Personal Relationships. 1995; 12(3): 463-472. doi:10.1177/0265407595123009
- [Background] Bonuck KA, Goodlin-Jones BL, Schechter C, Owens J. Modified Children's sleep habits questionnaire for behavioral sleep problems: A validation study. Sleep Health. 2017 Jun;3(3):136-141. doi: 10.1016/j.sleh.2017.03.009. Epub 2017 Apr 8. PMID 28526249
- [Background] Brooke J. System Usability Scale (SUS): A quick and dirty usability scale. Digital Equipment Corporation. 1986. Retrieved 1/2/18 from usability.gov website: https://www.usability.gov/how-to-andtools/methods/system-usability-scale.html
- [Background] Driscoll K, Pianta RC. Mothers' and fathers' perceptions of conflict and closeness in parent-child relationships during early childhood. Journal of Early Childhood and Infant Psychology. 2011; 7: 1-24.
- [Background] Louie AD, Cromer LD, Berry JO. Assessing parenting stress: Review of the use and interpretation of the Parental Stress Scale. The Family Journal, 2017; 25: 359-367. doi:10.1177/1066480717731347
- [Background] Morawska A, Sanders MR, Haslam D, Filus A, Fletcher R. Child Adjustment & Parent Efficacy Scales (CAPES): Development and initial validation of a parent-report measure. Australian Psychologist. 2014; 49: 241-252.
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Background] Sanders MR, Morawska A, Haslam DM, Filus A, Fletcher R. Parenting and Family Adjustment Scales (PAFAS): validation of a brief parent-report measure for use in assessment of parenting skills and family relationships. Child Psychiatry Hum Dev. 2014 Jun;45(3):255-72. doi: 10.1007/s10578-013-0397-3. PMID 23955254
- [Background] Zelman JJ, Ferro MA. The Parental Stress Scale: Psychometric properties in families of children with chronic health conditions. Family Relations. 2018; 67(2): 240-252.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | The Talk Parenting Skill for Alexa - Parent | The Talk Parenting Skill for Alexa - Child
Started | 49 | 49
Completed | 17 | 17
Not Completed | 32 | 32
Not completed — Lost to Follow-up | 32 | 32

BASELINE CHARACTERISTICS:
Population: Although the 49 children were considered enrolled participants that actively participate in the intervention, we obtained no assessment data from the children themselves. We do have basic demographic data as reported by the parent.
Groups:
- Total: Total of all reporting groups
Arm/Group | The Talk Parenting Skill for Alexa - Parent | The Talk Parenting Skill for Alexa - Child | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of the parent
  years | 34.4 (6.5) | 5.0 (0.8) | 19.7 (3.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 45 | 20 | 65
  Male | 1 | 27 | 28
  Non-binary | 1 | 0 | 1
  Unknown | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 43 | 41 | 84
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 3 | 5
  White | 38 | 36 | 74
  More than one race | 4 | 7 | 11
  Unknown or Not Reported | 3 | 3 | 6
Relationship Status [Count of Participants; unit: Participants] — The relationship status of the parent
  Participants
    Single, never married | 10 | 0 | 10
    Single, divorced | 5 | 0 | 5
    Unmarried, living with partner | 9 | 0 | 9
    Married | 20 | 0 | 20
    Married, separated | 3 | 0 | 3
    Unknown | 2 | 0 | 2
    Not Applicable | 0 | 49 | 49

OUTCOME MEASURES:

1. Primary Outcome: Parenting and Family Adjustment Scales (PAFAS): Positive Encouragement Subscale
Description: The Positive Encouragement and Coercive Parenting subscales of the Parenting and Family Adjustment Scales (PAFAS) are used to measure parents' positive encouragement and coercive parenting. The Positive Encouragement subscale is measured with three items, answered on a 4-point scale (0=Not at all; 3=Very much); summed scores range from 0 to 9, with higher scores indicating worse outcomes. The Coercive Parenting subscale is measured with five items, answered on the same 4-point scale; summed scores range from 0 to 15, with higher scores indicating worse outcomes. Each subscale shows good internal consistency and construct validity.
Time Frame: Baseline (T1), 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- The Talk Parenting Skill for Alexa: 49 parents will be assessed at enrollment, then provided an Amazon Echo Dot and exposed to the prototype Bedtime Routine module of the Talk Parenting program for 4 weeks, and then re-assessed at 4 weeks (at treatment completion)
  The Talk Parenting Skill for Alexa: In a 4-week period, families use at home a prototype Bedtime Routine module of the Talk Parenting program, a smart speaker app designed to provide parents with in-situ experiential support for building positive family routines. The prototype Bedtime Routine module of Talk Parenting guides families in creating a healthy bedtime routine to foster healthy sleep habits, provide experiential practice in self-regulation skills, and promote a positive parent-child relationship.
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale
  Pretest | 2.53 (2.12)
  Posttest | 2.76 (1.44)
Statistical Analysis 1: Comparison: The Talk Parenting Skill for Alexa; Test type: Equivalence — Test of whether the pretest and posttest scores are significantly different from zero; p = .690, t-test, 2 sided; Mean Difference (Final Values) = 0.23, Standard Error of Mean .56 — Estimation parameter based on paired t-test

2. Primary Outcome: Parenting and Family Adjustment Scales (PAFAS) - Coercive Parenting Subscale
Description: as for outcome 1
Time Frame: Baseline (T1), 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale
  Pretest | 3.53 (1.23)
  Posttest | 2.88 (1.54)
Statistical Analysis 1: Comparison: The Talk Parenting Skill for Alexa; Test type: Equivalence — Test of whether pretest to posttest score change is greater than zero; p = .052, t-test, 2 sided; Mean Difference (Final Values) = .647, Standard Error of Mean .308

3. Primary Outcome: Child Adjustment and Parent Self-Efficacy Scale (CAPES) - Emotional Adjustment Subscale
Description: The Child Adjustment and Parent Efficacy Scale (CAPES) measures children's behaviors and emotional adjustment. The Behavior Problems subscale consists of 16 problematic and 8 reverse-coded positive behaviors. Respondents answer on a 4-point scale (0=Not at all; 3=Very much); the summed scores range from 0 to 72, with higher scores indicating worse outcomes. The Emotional Maladjustment subscale has 3 items. Respondents answer on the same 4-point scale; the summed scores range from 0 to 9, with higher scores indicating worse outcomes. The CAPES is also used to measure parents' self-efficacy; parents rate their confidence that they can successfully deal with each of the 19 negative behaviors/emotions on the CAPES. Respondents answer on a 10-point scale (1=Certain I can't do it; 10=Certain I can do it); the summed scores range from 19-190, with higher scores indicating better outcomes.
Time Frame: Baseline (T1), 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale
  Pretest | 2.06 (2.70)
  Posttest | 1.41 (1.77)
Statistical Analysis 1: Comparison: The Talk Parenting Skill for Alexa; Test type: Equivalence — Test of whether pretest to posttest change is significantly different from zero; p = .135, t-test, 2 sided; Mean Difference (Final Values) = .647, Standard Error of Mean .410

4. Primary Outcome: Child Adjustment and Parent Self-Efficacy Scale (CAPES) - Behavior Problems Subscale
Description: as for outcome 3
Time Frame: Baseline (T1), 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale
  Pretest | 31.24 (10.23)
  Posttest | 27.00 (9.32)
Statistical Analysis 1: Comparison: The Talk Parenting Skill for Alexa; Test type: Equivalence — Test of whether pretest to posttest change is significantly different from zero; p = .026, t-test, 2 sided; Mean Difference (Final Values) = 4.24, Standard Error of Mean 7.14

5. Primary Outcome: Short-Form Children's Sleep Habits Questionnaire (SF-CSHQ)
Description: Children's bedtime/sleep problems is measured with the Short-Form Children's Sleep Habits Questionnaire (SF-CSHQ), a 23-item version of the widely used Children's Sleep Habits Questionnaire (CSHQ). Respondents answer on a 5-point scale (1=never; 5=always); average scores range from 1 to 5, with higher scores indicating worse outcomes. The SF-CSHQ shows good validity against the original CSHQ, external validity, internal reliability, and sensitivity to change.
Time Frame: Baseline (T1), 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale
  Pretest | 2.78 (0.46)
  Posttest | 2.30 (0.40)
Statistical Analysis 1: Comparison: The Talk Parenting Skill for Alexa; Test type: Equivalence — Test of whether pretest to posttest change is significantly different from zero; p < .001, t-test, 2 sided; Mean Difference (Final Values) = 0.48, Standard Error of Mean 0.09

6. Primary Outcome: Program-Targeted Parenting Practices - Frequency of Engagement Subscale
Description: Frequency of parents' engagement in the parenting practices targeted by the intervention, and parents' self-efficacy for doing so, are measured by the Program-Targeted Parenting Practices measure. Created by the Investigators, 14 items ask parents to report the frequency with which they have engaged in target parenting practices related to bedtime in the past 4 weeks, on a 6-point scale (0=Never in past month; 5=Every day in past month); average scores range from 0 to 5, higher scores indicating better outcomes. Then parents are asked to rate how confident they are in doing 12 of these target parenting practices, on a 10-point scale (1=Not at all confident; 10=Highly confident); average scores range from 1 to 10, higher scores indicating better outcomes. Finally, 3 items ask parents for their satisfaction with how child's bedtime is going, on a 10-point scale (0=Not at all satisfied; 10=Very satisfied); average scores range from 1 to 10, higher scores indicating better outcomes.
Time Frame: Baseline (T1), 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale
  Pretest | 3.40 (0.75)
  Posttest | 4.05 (0.48)
Statistical Analysis 1: Comparison: The Talk Parenting Skill for Alexa; Test type: Equivalence — Test of whether pretest to posttest change is significantly different from zero; p < .001, t-test, 2 sided; Mean Difference (Final Values) = -0.66, Standard Error of Mean 0.13

7. Primary Outcome: Program-Targeted Parenting Practices - Self-Efficacy of Practice Subscale
Description: as for outcome 6
Time Frame: Baseline (T1), 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale
  Pretest | 7.24 (2.46)
  Posttest | 8.35 (1.12)
Statistical Analysis 1: Comparison: The Talk Parenting Skill for Alexa; Test type: Equivalence — Test of whether pretest to posttest change is significantly different from zero; p = .057, t-test, 2 sided; Mean Difference (Final Values) = -1.11, Standard Error of Mean 0.54

8. Primary Outcome: Program-Targeted Parenting Practices - Satisfaction Handling Bedtime Subscale
Description: as for outcome 6
Time Frame: Baseline (T1), 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale
  Pretest | 4.18 (2.14)
  Posttest | 7.62 (1.44)
Statistical Analysis 1: Comparison: The Talk Parenting Skill for Alexa; Test type: Equivalence — Test of whether pretest to posttest change is significantly different from zero; p < .001, t-test, 2 sided; Mean Difference (Final Values) = -3.44, Standard Error of Mean 1.89

9. Primary Outcome: Child-Parent Relationship Scale - Short Form (CPRS) - Closeness Subscale
Description: The Child-Parent Relationship Scale - Short Form (CPRS-SF) is used to measure the degree of closeness and conflict in the parent-child relationship. The CPRS-SF is comprised of 15 parent-report items that ask the parent for their assessment of the child-parent relationship, the child's emotional stance toward the parent, and the parent's feelings toward the child. Two subscales are derived: Conflicts and Positive Aspects/Closeness. The Conflicts subscale is measured by 7 items on a 5-point scale (1=Definitely does not apply; 5=Definitely applies); average scores range from 1 to 5, with higher scores indicating worse outcomes. The Closeness subscale is measured with 7 items on the same 5-point scale; average scores range from 1 to 5, with higher scores indicating better outcomes. The CPRS-SF has been validated with parents of preschoolers and first graders and shows good internal consistency.
Time Frame: Baseline (T1), 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale
  Pretest | 4.74 (0.35)
  Posttest | 4.83 (0.18)
Statistical Analysis 1: Comparison: The Talk Parenting Skill for Alexa; Test type: Equivalence — Test of whether pretest to posttest change is significantly different from zero; p = .352, t-test, 2 sided; Mean Difference (Final Values) = -0.09, Standard Error of Mean 0.10

10. Primary Outcome: Child-Parent Relationship Scale - Short Form (CPRS) - Parent-Child Conflict Subscale
Description: as for outcome 9
Time Frame: Baseline (T1), 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale
  Pretest | 2.69 (0.69)
  Posttest | 2.46 (0.67)
Statistical Analysis 1: Comparison: The Talk Parenting Skill for Alexa; Test type: Equivalence — Test of whether pretest to posttest change is significantly different from zero; p = .104, t-test, 2 sided; Mean Difference (Final Values) = 0.23, Standard Error of Mean 0.13

11. Primary Outcome: System Usability Scale (SUS)
Description: Skill usability is measured with the System Usability Scale (SUS), a commonly used 10-item scale that measures subjective perceptions of usability. Items are answered on a 5-point scale (1=Strongly disagree; 5=Strongly agree). The value of one is subtracted from odd numbered items (1, 3, 5, 7, and 9) and the even number items (2, 4, 6, 8, and 10) are subtracted from the value of five. Scores are then summed and multiplied by 2.5 resulting in scores on a scale that ranges from 1 to 100, with higher scores indicating better usability.
Time Frame: At 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale | 78.8 (20.7)

12. Primary Outcome: Program Acceptability
Description: Program acceptability was measured with 7 items at T2, 4 weeks after baseline, asking the extent to which primary parents found the Talk Parenting skill useful, enjoyable, whether it addressed important topics, helped make bedtime more positive, enjoyment of use by child, how much use of bedtime strategies, and how much bedtime strategies helped the child and family. Respondents answer items on a 7-point scale (1=Not at all; 7=Very much); average scores range from 1 to 7, with higher scores indicating better satisfaction.
Time Frame: At 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale | 5.30 (1.50)

13. Secondary Outcome: Self-Efficacy for Parenting Tasks Index (SEPTI) - Toddler Scale - Discipline Subscale
Description: The Self-Efficacy for Parenting Tasks Index - Toddler Scale - Short Form (SEPTI-TS-SF) is used to measure parents' self-efficacy for a discipline- and routines-related parenting tasks. The Discipline and Routines subscales are measured with 6 items each. Respondents answer on a 6-point scale (1=Agree strongly; 6=Disagree strongly); average scores range from 1 to 6, with higher scores indicating better outcomes. These SEPTI-TS-SF subscales show good internal consistency, construct validity, and discriminant validity, and sensitivity to change.
Time Frame: Baseline (T1), 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale
  Pretest | 3.30 (1.18)
  Posttest | 3.64 (1.04)
Statistical Analysis 1: Comparison: The Talk Parenting Skill for Alexa; Test type: Equivalence — Test of whether pretest to posttest change is significantly different from zero; p = .106, t-test, 2 sided; Mean Difference (Final Values) = -0.33, Standard Error of Mean 0.19

14. Secondary Outcome: Self-Efficacy for Parenting Tasks Index (SEPTI) - Toddler Scale - Routine Subscale
Description: as for outcome 13
Time Frame: Baseline (T1), 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale
  Pretest | 4.18 (1.26)
  Posttest | 4.81 (0.88)
Statistical Analysis 1: Comparison: The Talk Parenting Skill for Alexa; Test type: Equivalence — Test of whether pretest to posttest change is significantly different from zero; p = .005, t-test, 2 sided; Mean Difference (Final Values) = -0.64, Standard Error of Mean 0.19

15. Secondary Outcome: Parental Stress Scale (PSS)
Description: The Parental Stress Scale (PSS) is used to measure parents' stress level. The PSS is comprised of 18 items that ask about positive (emotional benefits, personal development) and negative (demands on resources, restrictions) themes of parenthood. Respondents answer on a 5-point scale (1=Strongly disagree; 5=Strongly agree); summed scores range from 18 to 90, with higher scores indicating worse outcomes. The PSS shows good internal consistency, test-retest reliability, discriminant validity, and construct validity and has been validated across cultures and languages, with families of typically developing children, and with families of children with emotional/ behavioral problems, developmental disabilities, and chronic health conditions.
Time Frame: Baseline (T1), 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 17
units on a scale
  Pretest | 39.35 (6.24)
  Posttest | 35.82 (8.67)
Statistical Analysis 1: Comparison: The Talk Parenting Skill for Alexa; Test type: Equivalence — Test of whether pretest to posttest change is significantly different from zero; p = .082, t-test, 2 sided; Mean Difference (Final Values) = 3.52, Standard Error of Mean 1.90

16. Secondary Outcome: Families' Usage of the Talk Parenting (TP) Skill - Number of Families That Activated the Skill
Description: Families' usage of the TP skill is measured through usage metrics and transcripts collected on the back-end database, including number of families that activated the skill, number of times skill was used, number of steps a family used, length of bedtime routine in minutes, and number of families that listened to a podcast. Higher levels for all metrics indicate greater skill use.
Time Frame: At 4 weeks after baseline (T2)
Measure: Count of Participants; unit: Participants
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 27
Participants | 20

17. Secondary Outcome: Families' Usage of the Talk Parenting (TP) Skill - Number of Times Skill Was Used
Description: as for outcome 16
Time Frame: At 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: Number of times
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 20
Number of times | 15 (19.2)

18. Secondary Outcome: Families' Usage of the Talk Parenting (TP) Skill - Number of Steps Used
Description: as for outcome 16
Time Frame: At 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: Number of steps
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 20
Number of steps | 10.4 (2.8)

19. Secondary Outcome: Families' Usage of the Talk Parenting (TP) Skill - Length of Bedtime Routine
Description: as for outcome 16
Time Frame: At 4 weeks after baseline (T2)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 20
Minutes | 35.0 (19.2)

20. Secondary Outcome: Families' Usage of the Talk Parenting (TP) Skill - Listened to a Podcast
Description: as for outcome 16
Time Frame: At 4 weeks after baseline (T2)
Measure: Count of Participants; unit: Participants
Arm/Group | The Talk Parenting Skill for Alexa
Number analyzed (Participants) | 20
Participants | 12

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from completion assessment through the final 4-week posttest period.
Arm/Group | The Talk Parenting Skill for Alexa - Parent | The Talk Parenting Skill for Alexa - Child
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT04633434/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT04633434/ICF_001.pdf